CLINICAL TRIAL: NCT03303690
Title: A Prospective Trial on the Clinical Efficacy of the Ankle Spacer for the Surgical Treatment of Large, Multiple, Cystic and Secondary or Tertiary Osteochondral Defects of the Talus
Brief Title: AS: Ankle Spacer for Talar Osteochondral Defects
Acronym: AS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Arthrex stopped manufacturing the device
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Jari Dahmen, Local Study Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GK2017AS
Record Dates: First submitted 2017-09-17; First posted 2017-10-06 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Osteochondral Defect of Talus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ankle Spacer (AS) (Experimental): This arm will surgically receive the to be implanted ankle spacer in their ankle.
  Interventions: Procedure: Ankle Spacer (AS)

INTERVENTIONS:
Procedure: Ankle Spacer (AS) — All included patients will be treated by means of surgical implantation of the Ankle Spacer prosthesis in an open manner replacing the talar side of the tibiotalar joint.

SUMMARY:
By means of the Ankle Spacer patients will be implanted, the clinical and radiological results of which will be prospectively recorded and analyzed at different points in time.

DETAILED DESCRIPTION:
Ankle sprains can result in talar osteochondral defects (OCDs) which have a significant impact on the quality of life of patients. When these OCDs are of large nature (anterior-posterior or medial-lateral diameter >1.5cm in diameter), cystic, have failed prior surgical treatment, or when there are multiple present on the talar articular surface, surgical care by means of fixation or bone marrow stimulation is contra-indicated. An ankle arthrodesis or fusion can be considered, but this results in functional limitation due to a decreased range of motion (ROM). In order to serve for a bone sparing prosthesis procedure, preserve range of motion, optimize physical functioning and to resurface the talus, the Ankle Spacer has been developed. It is a one-piece implant system that replaces the articulating upper talus surface of the tibio-talar joint, and offers several implant sizes in order to fit to the different talus sizes. It is anatomically designed to the native upper talus surface to provide an optimal fit to the distal articular surface. It has a rough titanium plasma spray (TPS) coated under surface with two posts and spikes for implant fixation. The rough surface enables secondary fixation by means of bone ingrowth and the spikes at the posterior part of the prosthesis allowing for optimal adherence of the implant and for minimal iatrogenic damage upon fixation. By these means, the anatomical situation and the natural congruency of the ankle joint are mirrored to a optimal extent. Despite the fact that no clinical trials have been published on this specific implant, it is hypothesized that the 5-year postoperative clinical outcomes concerning pain and prosthesis survival will be considered good.

ELIGIBILITY:
Inclusion Criteria:

* age ranging from 18 to 80 years
* talar osteochondral defect (multiple degenerative talar cysts present, and/or prior failed surgical treatment and/or multiple defects and/or large (>15mm))
* willing to receive surgical implantation of the Ankle Spacer
* has been informed of the nature of the study and provided written consent
* The subject and treating physician agree that the subject will return for all required post-procedure follow-up visits
* failed previous conservative treatment
* complaints for at least 6 months

Exclusion Criteria:

* -severe ankle malalignement.(> 5° varus/valgus).
* fracture < 6 months - tendinitis - diabetes mellitus / rheumathoid arthritis
* advanced osteoporosis
* grade two or higher (Kellgren-Lawrence-Score) ankle joint degeneration on the tibia side.
* any ankle deformation that does not allow proper rasping of the cartilage and/or proper seating of the desired sized implant, as described in the surgical technique.
* blood supply limitations and previous infections, which may retard healing.
* foreign-body sensitivity. Where material sensitivity is suspected, appropriate tests should be made and sensitivity ruled out prior to implantation.
* active infection or blood supply limitations.
* conditions that tend to limit the patient's ability or willingness to restrict activities or follow directions during the healing period, including severe neuro-arthropathy.
* pathological conditions, such as insufficient quantity or quality of bone (e.g., cystic changes or severe osteopenia), which may compromise implant fixation.
* currently participating in an investigational drug or another device study that clinically interferes with the current study endpoints.
* Inability to be brought back to the surgery site for long term follow-up evaluations or the subject is unwilling to fill out the appropriate evaluation forms
* adiposity grade I (BMI > 30 kg/m2)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-12-05 (Actual); Primary Completion 2020-03-11 (Actual); Study Completion 2020-03-11 (Actual)

PRIMARY OUTCOMES:
NRS during walking/weightbearing | 2 years postoperatively
  The primary study parameter is the measurement of the NRS

SECONDARY OUTCOMES:
NRS at rest and during stairclimbing | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other outcome measures will include pain evaluation using the NRS pain at rest and during stair climbing
NRS during stairclimbing | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other outcome measures will include pain evaluation using the NRS pain at rest and during stair climbing
AOFAS (American Orthopedic Foot and Ankle Score) | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other outcome measures will include the AOFAS.
FAOS (Foot and Ankle Outcome Score) | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other outcome measures will include FAOS
SF-36 (Short-Form 36) Physical Component Scale | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other outcome measures will include SF-36 Physical Component Scale
SF-36 (Short-Form 36) Mental Component Scale | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other outcome measures will include SF-36 Mental Component Scale
ROM (range of motion) | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other outcome measures will include Range of Motion (ROM) in degrees of dorsi- and plantarflexion and will be measured using a goniometer
demographic data: sex | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other study parameters that will be recorded are demographic data and also radiographic evaluations to evaluate loosening and subsidence (radiographs). Complications, implant survivorship (revision rate), operation time, adverse events, and length of hospital stay will also be recorded.
demographic data: age | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Other study parameters that will be recorded are demographic data and also radiographic evaluations to evaluate loosening and subsidence (radiographs). Complications, implant survivorship (revision rate), operation time, adverse events, and length of hospital stay will also be recorded.
Radiographic evaluation | pre-operatively, follow-ups at 2 weeks, 6 weeks, 3 months, 6 months, 1,2,3,4,5 year postop.
  Radiographic evaluations to evaluate loosening and subsidence (radiographs). Complications, implant survivorship (revision rate), operation time, adverse events, and length of hospital stay will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: G.M.M.J. Kerkhoffs, MD PhD, Principal Investigator — Academic Medical Center (AMC Amsterdam)
Locations (1):
- Academic Medical Center, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No